# **Study Protocol**

Title: The Impact of Robot-assisted Digital Education on Prenatal Women's Health Literacy

NCT Number: NCT20230940

Document Date: 2025-05-04

### 1. Background and Rationale

The study addresses the increasing need for efficient, standardized prenatal health education, especially in light of nursing workforce shortages. Robot-assisted education presents a novel digital solution that may reduce anxiety and enhance health literacy among pregnant women, particularly those diagnosed with gestational diabetes mellitus (GDM).

## 2. Study Objectives

- Primary Objective: To evaluate whether robot-assisted digital education reduces anxiety among pregnant women with GDM.
- Secondary Objectives: To examine the impact on health literacy, satisfaction with health education, and acceptance of digital technologies.

## 3. Study Design

Type: Randomized Controlled Trial (RCT)

Setting: Obstetrics outpatient clinic of a regional hospital in Taiwan

Duration: November 2023 to January 2024

Groups:

- Experimental group: Robot-assisted education - Control group: Tablet-based video education Blinding: Single-blind (participant and assessor)

## 4. Participants

**Inclusion Criteria:** 

- Pregnant women aged ≥21
- GDM diagnosis
- Taiwanese nationality

**Exclusion Criteria:** 

- Chronic illness
- Cognitive impairment or language barrier

#### 5. Intervention

A 30-minute robot-assisted session on GDM information using visual, audio, and interactive storytelling features.

#### 6. Outcomes

Primary: Hamilton Anxiety Rating Scale (HAMA)

Secondary: Health Literacy Questionnaire (HLQ), Satisfaction (adapted Black et al.),

**Technology Acceptance** 

#### 7. Ethics

Approved by the Institutional Review Board of Taipei Medical University. Informed consent obtained(ethical approval number N202309040).

## 8. Data Availability

Available upon reasonable request to the corresponding author.

# Statistical Analysis Plan

Title: Statistical Analysis Plan for the RCT "The Impact of Robot-assisted Digital Education on Prenatal Women's Health Literacy"

NCT Number: NCT20230940

Document Date: 2025-05-04

## 1. Sample Size Calculation

Using G\*Power with a medium effect size (d = 0.5), alpha = 0.05, power = 0.80. Minimum of 64 participants required. Target recruitment: 80 (to allow for dropouts).

#### 2. Randomization

Block randomization via computer-generated sequence. Allocation concealed until participant assignment.

### 3. Analysis Methods

Baseline Characteristics: Independent t-tests or chi-square Primary Outcome (Anxiety): Independent samples t-test Secondary Outcomes:

- Health literacy, satisfaction, technology acceptance: t-tests
- Associations: One-way ANOVA and chi-square tests

Software Used: SPSS v25

Missing Data: Excluded from per-protocol; ITT analysis with multiple imputation

recommended in future studies

## 4. Significance Level

Two-tailed tests with  $\alpha = 0.05$ .